CLINICAL TRIAL: NCT01410552
Title: Inappropriate Shock Reduction wIth PARAD+ Rhythm DiScrimination
Acronym: ISIS-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS ICD - ITSY09
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Tachycardia
Keywords: Primary prevention; Secondary prevention
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Intervention Model Description: ICD device

ARMS (1):
- ICD or CRT-D with PARAD+ (Other): only 1 arm is the study: all patients implanted with ICD or CRT-D with PARAD+ enabled, no comparator
  Interventions: Device: PARADYM DR model 8550; PARADYM CRT model 8750; PARADYM RF DR model 9550; PARADYM RF CRT model 9750; PARADYM RF CRT SonR model 9770

INTERVENTIONS:
Device: PARADYM DR model 8550; PARADYM CRT model 8750; PARADYM RF DR model 9550; PARADYM RF CRT model 9750; PARADYM RF CRT SonR model 9770 — PARADYM ICD and CRT-d with PARAD+ algorithm available

SUMMARY:
ISIS- ICD study has been designed to evaluate the impact of PARAD+ algorithm on inappropriate shocks, in a general population implanted for primary or secondary prevention with a dual or tri chamber device at one year follow-up

DETAILED DESCRIPTION:
The primary endpoint is to demonstrate that 95% of patients implanted with PARAD+ algorithm are free from inapproporiate shock compared to 92.5% in general ICD population.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible for implantation (according to current accepted guidelines, or scheduled for implant (primo-implant, replacement, upgrade) with a Paradym/Paradym RF (CRT-D or DR-ICD) within the next 30 days, or has already been implanted within the last 30 days
2. Patient in sinus rhythm, or patients with paroxysmal atrial tachyarrhythmia or patients with persistent atrial tachyarrhythmia in whom a cardioversion is planned within three months

Exclusion Criteria:

1. Any contraindication for ICD therapy
2. Atrial lead not implanted
3. Patient with permanent atrial tachyarrhythmia
4. Patients implanted with a ventricular assist device (VAD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo RUIZ GRANELL, Dr, Principal Investigator — Cardiology Department Arrhythmia Unit Hospital Clinico Universitario Valencia SPAIN; Mark RICHARDS, Dr., Principal Investigator — Toledo Hospital, 4614 Brookside Dr. Toledo (OH)
Locations (80):
- United States (27):
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Pacific Arrhythmia Services, Mesa, Arizona
  - Banner Arizona Medical Clinic, Peoria, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Southern California Electrophysiology Associates, Anaheim, California
  - Raymond H. M. Schaerf MD, Inc., Burbank, California
  - St. Rose Hospital, Fremont, California
  - H. Raj Reddy Md, Inc., Hanford, California
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial West Hospital, Pembroke Pines, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - University of Chicago, Chicago, Illinois
  - St. Tammany Hospital, Covington, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - MGH, Boston, Massachusetts
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Harlem Cardiology, New York, New York
  - Pitt Memeorial Hospital Heart Rhythm Associates, Greenville, North Carolina
  - Rex Heart and Vascular Specialists, Raleigh, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Easton Hospital, Easton, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Providence Hospital, Columbia, South Carolina
  - Carolina Arrhythmia Consultants, Mt. Pleasant, South Carolina
- France (22):
  - Centre Hospitalier Universitaire D'Amiens, Amiens
  - Clinique Saint Joseph, Angers
  - Chu Annecy, Annecy
  - CH Henri Duffaut - Avignon, Avignon
  - Hôpital Privé de Bois Bernad, Bois-Bernard
  - CHRU du Morvan Hôpital la Cavale Blanche, Brest
  - Hôpital Instruction des Armées, Clamart
  - CH La Rochelle - hôpital St Louis, La Rochelle
  - CH LENS, Lens
  - Hopital Saint Joseph et saint Luc, Lyon
  - Centre Hospitalier Universitaire de La Timone, Marseille
  - Hopital Nord, Marseille
  - CH Montpellier, Montpellier
  - CH Emile Muller, Mulhouse
  - CHU Groupe Hospitalo-universitaire Caremeau, Nîmes
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier, Pau
  - CH Périgueux, Périgueux
  - CH Yves le Foll, Saint-Brieuc
  - Centre Hospitalier de Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Klinikum Bogenhausen, Bogenhausen
  - Universitatsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - UKSH Campus Luebeck, Lübeck
  - Klinik für Kardiologie Städtisches Klinikum Lüneburg gGmbH, Lüneburg
  - Kardiologische Praxis Dr. med Taggeselle, Markkleeberg
  - DRK Krankenhaus Ratzeburg, Ratzeburg
- Italy (3):
  - Policlinico Consorziale di Bari U.O Cardiologia Universitaria, Bari
  - Po Melorio, Santa Maria Capua Vetere
  - Ospedale S.Andrea, Vercelli
- Japan (13):
  - Chiba University Hospital, Chiba
  - Ichinomiya Nishi Hospital, Ichinomiya
  - Iizuka Hospital, Iizuka
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kokura Memorial Hospital, Kokura
  - Ohtanishinouchi Hospital, Kōriyama
  - Shin-Tokyo Hospital, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Tokyo Metropolitan Hiroo Hospital, Tokyo
  - Tokai University School of Medicine, Tōkai
  - Yamaguchi University Hospital, Ube
  - Yokohama City University Hospital, Yokohama
  - Yokohama Rosai general Hospital, Yokosuka
- Spain (4):
  - Hospital Universitario de la Ribera, Alzira
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario La Paz, Madrid
  - CHU VIGO, Vigo
- United Kingdom (5):
  - Basildon University Hospital, Basildon, England
  - Blackpool Victoria Hospital, Blackpool
  - Papworth Everard, Cambridge
  - Dorset County Hospital, Dorchester
  - Kettering Hospital, Kettering

REFERENCES:
- [Derived] Ruiz-Granell R, Dovellini EV, Dompnier A, Khalighi K, Garcia-Campo E, Olivier A, Barcelo A, Ritter P. Algorithm-based reduction of inappropriate defibrillator shock: Results of the Inappropriate Shock Reduction wIth PARAD+ Rhythm DiScrimination-Implantable Cardioverter Defibrillator Study. Heart Rhythm. 2019 Sep;16(9):1429-1435. doi: 10.1016/j.hrthm.2019.03.016. Epub 2019 Mar 22. PMID 30910709

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICD or CRT-D With PARAD+
Started | 1013
Completed | 877
Not Completed | 136

BASELINE CHARACTERISTICS:
Population: The PARAD+ algorithm was enabled in implanted devices in 993 subjects, 639 with an ICD and 354 with a CRT-D, who were thus considered for the primary analysis.
Groups:
- Single Arm: ICD or CRT-D with PARAD+
Arm/Group | Single Arm
Number analyzed (Participants) | 993
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.0 [60.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 789
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patients With Inappropriate Shock(s)
Description: Percentage of patients presenting with inappropriate shock(s)
Time Frame: 552 days
Measure: Number; unit: Percentage of pts with inap shocks
Arm/Group | Single Arm
Number analyzed (Participants) | 993
Percentage of pts with inap shocks | 1.4

2. Secondary Outcome: Shock(s) Appropriately Delivered
Description: Percentage of shocks appropriately delivered
Time Frame: 552 days
Measure: Number; unit: Percentage of appropriate shocks
Arm/Group | Single Arm
Number analyzed (Participants) | 993
Percentage of appropriate shocks | 73.7

ADVERSE EVENTS:
Time Frame: Over a median follow up of 552 days (Q1: 354.0; Q3: 725.0).
Description: Serious adverse events and hospitalizations were documented on specific case report forms and classified by the sponsor's safety officer.
  Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | ICD or CRT-D With PARAD+
All-Cause Mortality (participants affected / at risk) | 70/1013
Serious Adverse Events (participants affected / at risk) | 282/1013
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICD or CRT-D With PARAD+ (N=1013)
Cardiovascular serious adverse event (Cardiac disorders) | 165
Non cardiovascular serious adverse event (Respiratory, thoracic and mediastinal disorders) | 140
Device related serious adverse event (Investigations) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No